CLINICAL TRIAL: NCT05965323
Title: Reopening Schools Safely and Educating Youth Research- Early Learning Ancillary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Linda Ko, Professor, School of Public Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00014531-B; 1OT2HD107544-01 (NIH)
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Absenteeism
Keywords: SARS-coV-2; School re-opening; Rural Communities; Early Education - pre School; Risk communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The students in this arm will receive comic books and their parents videos on the benefits of preventive measures of COVID-19
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — Health education with comic books and videos

SUMMARY:
This is a single arm, pre/post intervention study to a larger trial that will examine the effect of health education with comic books and videos on COVID-19 preventive behaviors (masking, social distancing, testing and vaccine uptake). The participants are students, ages 3-5 years old and their parents.

DETAILED DESCRIPTION:
This is a single arm, pre/post intervention study to a larger trial that will examine the effect of health education with comic books and videos on COVID-19 preventive behaviors (masking, social distancing, testing and vaccine uptake). The participants are students, ages 3-5 years old and their parents.

Students will receive the intervention from November 2023 to March 2024.

ELIGIBILITY:
Inclusion Criteria:

* Must have a child attending the Early Learning Program in the Yakima School District
* Must be able to provide informed consent and legal guardian assent either virtually, on the telephone, or in-person.
* Must have a permanent mailing address available for study staff to mail necessary materials OR a working email address.
* Must speak English or Spanish.

Exclusion Criteria:

- Not in Early Learning program in Yakima School District

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ko, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of parent, child dyads in Early Learning anxillary study 09/22/2022 through 12/30/2022
Groups:
- Students: Assented students enrolled in Early Learning study
- Parent: Consented parents of Early Learning Students
Period: Overall Study
Arm/Group | Students | Parent
Started | 49 | 48
Completed | 49 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Recruitment of Early Learning students (3, 4 and 5 years old) and their parent or Guardian(s) regardless of their participation in SARS-CoV-2 testing provided by the Yakima School District.
Groups:
- Single Arm Pre and Post Intervention Study: We want to learn if health education (COVID-19 Health Education Comic Books and Videos) can increase the uptake of COVID-19 mitigation measures, improve children's school attendance, and increase families' physical and mental well-being using single-arm pre/post-study.
Arm/Group | Single Arm Pre and Post Intervention Study
Number analyzed (Participants) | 97
Age, Customized [Count of Participants; unit: Participants] — Population: Parent (n=48), Child (n=49) dyads, totaling (n=97) enrolled participants
  Participants
    Student: number analyzed (Participants) | 49
    Student: <18 years | 49
    Student: Between 18 and 65 years | 0
    Student: >65 years | 0
    Student: Unknown not reported | 0
    Parent: number analyzed (Participants) | 48
    Parent: <18 years | 0
    Parent: Between 18 and 65 years | 0
    Parent: >65 years | 0
    Parent: Unknown not reported | 48
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Parent (n=48), Child (n=49) dyads, totaling (n=97) enrolled participants
  Participants
    Student: number analyzed (Participants) | 49
    Student: Female | 23
    Student: Male | 26
    Student: Unknown, Not Reported | 0
    Parent: number analyzed (Participants) | 48
    Parent: Female | 36
    Parent: Male | 6
    Parent: Unknown, Not Reported | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Parent (n=48), Child (n=49) dyads, totaling (n=97) enrolled participants
  Participants
    Student: number analyzed (Participants) | 49
    Student: Hispanic or Latino | 40
    Student: Not Hispanic or Latino | 8
    Student: Unknown or Not Reported | 1
    Parent: number analyzed (Participants) | 48
    Parent: Hispanic or Latino | 34
    Parent: Not Hispanic or Latino | 8
    Parent: Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Parent (n=48), Child (n=49) dyads, totaling (n=97) enrolled participants
  Participants
    Student: number analyzed (Participants) | 49
    Student: American Indian or Alaska Native | 0
    Student: Asian | 0
    Student: Native Hawaiian or Other Pacific Islander | 0
    Student: Black or African American | 1
    Student: White | 8
    Student: More than one race | 0
    Student: Unknown or Not Reported | 40
    Parent: number analyzed (Participants) | 48
    Parent: American Indian or Alaska Native | 0
    Parent: Asian | 0
    Parent: Native Hawaiian or Other Pacific Islander | 0
    Parent: Black or African American | 1
    Parent: White | 7
    Parent: More than one race | 0
    Parent: Unknown or Not Reported | 40
Region of Enrollment [Number; unit: Student Participants]
  United States | 49
Region of Enrollment [Number; unit: Parent Participants] — Parent (n=48), Child (n=49) dyads, totaling (n=97) enrolled participants
  Parent Participants
    United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Testing
Description: Percentage of early learning students testing for COVID-19
Time Frame: Up to eleven months
Population: Early Learning Students age 3-5 years old
Measure: Count of Participants; unit: Participants
Groups:
- Early Learning: The students will receive comic books and their parents videos on the benefits of preventive measures of COVID-19
  Health Education: Health education with comic books and videos
Arm/Group | Early Learning
Number analyzed (Participants) | 49
Participants
  Enrollment: Test Yes | 41
  Enrollment: Testing No | 8
  Enrollment: Prefer not to Respond | 0
  Enrollment: Unknown Not Reported | 0
  Follow Up: Test Yes | 22
  Follow Up: Testing No | 20
  Follow Up: Prefer not to Respond | 1
  Follow Up: Unknown Not Reported | 6

2. Primary Outcome: Masking
Description: Percentage of early learning students masking for COVID-19
Time Frame: Up to eleven months
Population: Early Learning Students age 3-5 years old
Measure: Count of Participants; unit: Participants
Arm/Group | Early Learning
Number analyzed (Participants) | 49
Participants
  Enrollment: Frequently | 7
  Enrollment: Never | 21
  Enrollment: Sometimes | 21
  Enrollment: Missing | 0
  Follow Up: Frequently | 21
  Follow Up: Never | 15
  Follow Up: Sometimes | 7
  Follow Up: Missing | 6

3. Primary Outcome: Wash Hands
Description: Percentage of early learning students washing hands for COVID-19
Time Frame: Up to eleven months
Population: Early Learning Students age 3-5 years old
Measure: Count of Participants; unit: Participants
Arm/Group | Early Learning
Number analyzed (Participants) | 49
Participants
  Enrollment: Frequenty | 42
  Enrollment: Sometimes | 7
  Enrollment: Missing | 0
  Follow Up: Frequenty | 35
  Follow Up: Sometimes | 8
  Follow Up: Missing | 6

4. Primary Outcome: Hide Cough
Description: Percentage of early learning students who hide cough during COVID-19
Time Frame: Up to eleven months
Population: Early Learning Students age 3-5 years old
Measure: Count of Participants; unit: Participants
Arm/Group | Early Learning
Number analyzed (Participants) | 49
Participants
  Enrollment: Frequently | 13
  Enrollment: Sometimes | 24
  Enrollment: Never | 7
  Enrollment: Prefer not to Answer | 1
  Enrollment: Missing | 4
  Follow Up: Frequently | 14
  Follow Up: Sometimes | 24
  Follow Up: Never | 5
  Follow Up: Prefer not to Answer | 0
  Follow Up: Missing | 6

ADVERSE EVENTS:
Time Frame: Parent,(n=48), student (n=49) dyads were enrolled from 9/22/22 through 2/16/24.Adverse events were monitored for 1 year 5 months from baseline assessment through Post Survey.
Description: Definition is any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Single Arm Pre and Post Intervention Study - Parent; Single Arm Pre and Post Intervention Study - Child: We want to learn if health education (COVID-19 Health Education Comic Books and Videos) can increase the uptake of COVID-19 mitigation measures, improve children's school attendance, and increase families' physical and mental well-being using single-arm pre/post-study.
Arm/Group | Single Arm Pre and Post Intervention Study - Parent | Single Arm Pre and Post Intervention Study - Child
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 0/48 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT05965323/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05965323/SAP_001.pdf